CLINICAL TRIAL: NCT06493994
Title: Myval TransAXillary Transcatheter Aortic Valve Replacement Multicenter Clinical Registry
Acronym: MYVAL-TAX-TAVR
Status: Recruiting | Type: Observational
Sponsor: University of Luebeck (Other)
Collaborators: University Hopsital Schleswig Holstein Campus Lübeck (Other)
Responsible Party: Principal Investigator, Prof. Dr. med. Ingo Eitel, Head of the MKII, University of Luebeck
Other Study IDs: 2024-240
Record Dates: First submitted 2024-07-02; First posted 2024-07-10 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2025-01

CONDITIONS: Aortic Valve Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis | interventions — Taxes; Transcatheter Aortic Valve Replacement

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: transaxillary (TAX) transcatheter aortic valve replacement — Study goal is to determine the feasibility, procedural success, safety and potential benefit of the Myval transcatheter heart valve (THV) in patients undergone transaxillary (TAX) transcatheter aortic valve replacement (TAVR).

SUMMARY:
Study goal is to determine the feasibility, procedural success, safety and potential benefit of the Myval transcatheter heart valve (THV) in patients undergone transaxillary (TAX) transcatheter aortic valve replacement (TAVR).

ELIGIBILITY:
Inclusion Criteria:

* Patient has been treatet transaxillary (TAX) with Myval transcatheter aortic valve replacement
* BMI <35 kg/m2
* Ability to give informed consent

Exclusion Criteria:

* History of coronary artery bypass graft and a patent left internal mammary artery (LIMA)
* Age ≤18 years
* Patients presenting with pregnancy
* Patients without informed consent
* Expected life expectancy <2 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were treated with Myval TAVR via TAX access are included in the registry.
  The participating centers also provide a retrospective cohort of TAX-TAVR implantations with other TAVR prothesis (e.g. Edwards Sapien XT/3/Ultra, Medtronic Evolut R/Pro, Accurate Neo, Allegra, Portico) to compare the results and outcomes of the MYVAL-TAX-TAVR registry using the Myval THV with other TAVR bioprothesis used for TAX-TAVR. To further improve comparability between groups propensity score matching between the groups will be performed using the following parameters (age, sex, STS score, peripheral artery disease, atrial fibrillation, minimum axillary diameter, moderate/severe axillary tortuosity and moderate/severe axillary, calcification).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Time until first occurrence | 30 Days
  * Stroke including ischemic or hemorrhagic stroke,
  * Systemic embolism,
  * Major bleeding (BARC type 3-5), or Cardiovascular or unexplained death

CONTACTS AND LOCATIONS:
Locations (1):
- Universität zu Lübeck, Lübeck, Schleswig-Holstein, Germany

IPD SHARING:
Plan to Share IPD: No